CLINICAL TRIAL: NCT01388933
Title: A Multicenter, Randomized, Double-Blinded, Placebo-Controlled Study of Daikenchuto (TU-100) in Subjects With Moderate Crohn's Disease
Brief Title: A Safety and Efficacy Study of Daikenchuto (TU-100) to Treat Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to low enrollment
Sponsor: Tsumura USA (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TU100P2T2
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; natural; herbal; Kampo; inflammatory bowel disease; Adult ages 18 to 75; Male and female subjects
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — 12,13-dihydro-N-methyl-6,11,13-trioxo-5H-benzo(4,5)cyclohepta(1,2-b)naphthalen-5,12-imine; dai-kenchu-to

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TU-100 (Experimental): 15g TU-100 (oral, daily) for 8 consecutive weeks (administered as 5g three times daily)
  Interventions: Drug: TU-100
- Matching placebo (Placebo Comparator): Matching placebo given 5g three times daily orally for 8 consecutive weeks
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: TU-100 — 15g daily, orally as 5g three times daily for 8 consecutive weeks
  Other Names: Daikenchuto
  Arms: TU-100
Drug: Matching Placebo — 15g as 5g three times daily, orally for 8 consecutive weeks
  Other Names: Placebo
  Arms: Matching placebo

SUMMARY:
The purpose of this study is to determine whether Daikenchuto(TU-100)is effective in the treatment of Crohn's disease.

DETAILED DESCRIPTION:
Crohn's disease, a chronic condition resulting in inflammation of the gastrointestinal tract (GI), causes a person to experience persistent symptoms of inflammatory bowel disease, including abdominal pain, nausea, vomiting, rectal bleeding, diarrhea, and constipation, with infrequent bowel movements that are at times accompanied by a sensation of incomplete emptying after having a bowel movement. Tsumura's TU-100 is a modern herbal product that has been approved as a prescription drug in Japan. Several lines of evidence indicate that TU-100 attenuates intestinal inflammation in Crohn's disease by increasing intestinal blood flow and stimulating a protective lining of intestinal mucus which produces an anti-inflammatory effect. TU-100 may attenuate pathological changes in the intestine and reduce symptoms in patients with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* provide written informed consent
* ability to orally ingest study medication
* male or female between 18 to 75 inclusive
* diagnosed with Crohn's disease for at least 3 months
* CDAI score of 220-300 at screening
* sexually active participants of childbearing potential must agree to birth control
* no clinically significant conditions which the doctor would feel exclusionary
* stable medication (including probiotics)

Exclusion Criteria:

* history of any bowel condition that may interfere with the evaluation of the study drug
* positive stool cultures
* currently pregnant or lactating
* receiving total parenteral nutrition
* history of alcohol or drug abuse within one year
* history of malignancy within 5 years
* current use of anticholinergic agents, antidepressants during the study, warfarin, prokinetics, antipsychotic agents or narcotic analgesics
* treatment with Anti-TNF agents 12 weeks before screening
* treatment with corticosteroids four weeks prior to screening
* treatment with cyclosporine or tacrolimus eight weeks prior to screening
* presence of a poorly controlled medical condition
* history of allergic reaction to ginseng, ginger or sichuan pepper
* any use of supplemental ginger, ginseng and Sichuan powder 2 weeks prior to and through course of the trial
* current use of any of the following herbal medications: Boswellia, Cat's claw (Uncaria tomentosa), Cayenne pepper, Echinacea, Horsetail (Equisetum), Hops, Lady's mantle (Alchemilla), Marshmallow root (Althaea), Slippery elm (Ulmus rubra) Turmeric and White Willow (Salix alba)
* history of celiac disease
* current diagnosis of lactose intolerance
* history of any other investigational medication within 30 days of enrolling in study
* unsuitability as determined by the study doctor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Clinical response as measured by a reduction in the CDAI total score | over eight weeks

SECONDARY OUTCOMES:
CDAI reduction by number of points and difference from baseline | over eight weeks
proportion of subjects showing a clinical remission by measure of CDAI score | over eight weeks
The change in total CDAI score | every four weeks over eight weeks
The change in IBDQ total score and category sub-scores | every four weeks over eight weeks
The change in CRP level | every four weeks over eight weeks
The change in fecal calprotectin levels | over eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shunji Mochida, Ph.D., Study Director — Tsumura USA
Locations (27):
- United States (27):
  - Preferred Research Partners Inc, Little Rock, Arkansas
  - TRIMED Clinical Trials, Corona, California
  - Digestive Care Associates, LLC, San Carlos, California
  - University of California at San Francisco, San Francisco, California
  - Rocky Mountain Gastroenterology Associates, Lakewood, Colorado
  - Clinical Research of West Florida, Inc, Clearwater, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - University of Chicago Hospital Medical Center, Chicago, Illinois
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Metropolitan Gastroenterology Group. PC, Chevy Chase, Maryland
  - Endoscopic Microsurgery Associates PA, Towson, Maryland
  - MedRACS, Quincy, Massachusetts
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Digestive Health Center, Ocean Springs, Mississippi
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - NY Scientific CORP, Hollis, New York
  - PMG Research of Salisbury, Salisbury, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Ohio Gastroenterology and Liver, Cincinnati, Ohio
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Advanced Research Institute, Ogden, Utah
  - University of Washington Medical Center, Seattle, Washington